**Title of the Study**: Decision Making Study **Principal Investigator**: Mary A. Gerend, PhD

Florida State University College of Medicine

# What should I know about being in a research study?

• Whether or not you take part is up to you.

• You can choose not to take part.

- You can agree to take part and later change your mind.
- Your decision will not be held against you.
- You can ask all the questions you want before you decide.

# Why is this study being done?

The purpose of the study is to understand psychological factors that affect how people make decisions. To avoid influencing your participation or the study results, this consent form does not include complete information about the study hypotheses and the research questions being tested. You will be fully debriefed following your participation in the study.

### What will happen if I take part in this research study?

If you volunteer to be in this study, you will be asked to:

- Fill out a survey online
- Visit our lab at Florida State University (FSU) one time

The online survey will ask about your demographic characteristics, personality traits, health history, and previous experiences.

During the lab visit, the researcher may ask you to do the following:

- Record a short video to introduce yourself
- Watch and rate other videos
- Taste and rate some foods
- Complete short computer-based tasks
- Have your height, shape, and weight measured
- Provide three saliva samples
- Fill out surveys on your thoughts and emotions

# How long will the research last?

We expect that you will be in this study for a total of 135-140 minutes. The online survey should take about 15-20 minutes to complete. About one week later, you will be scheduled for a lab visit that is expected to take about 120 minutes.

# Is there any way being in this study could be bad for me?

- You may feel uncomfortable answering questions on the online survey or during the lab visit.
- You may feel uncomfortable or experience emotional distress when performing one or more of the study tasks.
- You may feel awkward when providing the saliva samples.

# Will being in this study help me in any way?

You will not directly benefit from your participation in the research. We cannot promise any benefits to others from your taking part in this research. However, the results of the research may benefit both the field of psychology as well as society, including the contribution to our deepened understanding about how we behave.

# What happens if I do not want to be in this research?

Participation in research is completely voluntary. You can decide to participate or not to participate. There are no alternatives to study participation. The alternative is to not participate in the study.

### How many people will be studied?

We expect about 320 people will be in this study.

### What are my responsibilities if I take part in this research?

If you take part in this research, you will be responsible for following these instructions to prepare for your lab visit. In the 1 hour before your lab visit:

- Do not eat any food or drink any beverages. (It is okay to drink water.)
- Do not smoke cigarettes or use e-cigarettes
- Do not exercise

Participants will take part in a food tasting and rating exercise during the lab visit. If you have an allergy to any of these ingredients (i.e., soybeans and its derivatives, wheat and its derivatives, gluten, milk, peanuts, tree nuts, potatoes, and/or eggs), please tell a member of the study team right away because the foods you will be tasting during the study contain these ingredients.

# What happens if I say "yes," but I change my mind later?

You do not have to take part in this study, but if you do, you can leave the research at any time, and it will not be held against you. Your decision whether to participate will not affect your relationship with Florida State University. You have the right to choose not to participate in any study activity or completely withdraw from continued participation at any point in this study without penalty to which you are otherwise entitled.

If you withdraw from the study, the researcher will ask you if the information/data/samples already collected can be used or whether they should be destroyed.

# What happens to the information collected for the research?

Any information that is obtained in connection with this study and that can identify you will remain confidential. It will be disclosed only with your permission or as required by law. None of your responses will be labeled with your name or any other identifiable information. You will be assigned a random unique identifier (ID number) that will be stripped of all personal information to protect confidentiality. Your responses to surveys and your saliva samples will be labeled with your ID number, but no information that could be linked back to you in any way. Access to the "key" linking personally identifiable information to your ID number will be restricted to the PI (Dr. Gerend). The "key" linking personally identifiable information to the participant ID numbers in the data set will be destroyed at the end of the research project. Reports will not identify individual participants and will use aggregated data. Dr. Gerend will oversee the data storage and reporting procedures. De-identified data will be stored into perpetuity.

The saliva samples you provide will be identified by ID number only. We will store your samples in a locked lab until they are processed. Samples will be analyzed for cortisol. After analysis has been completed, any remaining samples will be destroyed.

There are no plans to provide clinically relevant research results to you in this study.

Efforts will be made to limit the use and disclosure of your personal information, including research study data, to people who have a need to review this information. We cannot promise complete secrecy. Organizations that may inspect and copy your information include the IRB and other representatives of this organization.

When the study has ended, we will post the data on the Open Science Framework, which is a place where scientists share their data with other scientists and the public. However, this data will never include any of your personal information and will not include your name or any identifiable information.

This research is covered by a Certificate of Confidentiality from the National Institutes of Health. This means that the researchers cannot release or use information, documents, or samples that may identify you in any action or suit unless you say it is okay. They also cannot provide them as evidence unless you have agreed. This protection includes federal, state, or local civil, criminal, administrative, legislative, or other proceedings. An example would be a court subpoena.

There are some important things that you need to know. The Certificate DOES NOT stop reporting that federal, state, or local laws require. Some examples are laws that require reporting of child or elder abuse, some communicable diseases, and threats to harm yourself or others. The Certificate CANNOT BE USED to stop a sponsoring United States federal or state government agency from checking records or evaluating programs. The Certificate DOES NOT stop disclosures required by the federal Food and Drug Administration (FDA). The Certificate also DOES NOT prevent your information from being used for other research if allowed by federal regulations.

Researchers may release information about you when you say it is okay. For example, you may give them permission to release information to insurers, medical providers, or any other persons not connected with the research. The Certificate of Confidentiality does not stop you from willingly releasing information about your involvement in this research. It also does not prevent you from having access to your own information.

If identifiers are removed from your identifiable private information that is collected during this research, that de-identified information could be used for future research studies or distributed to another investigator for future research studies without your additional informed consent.

We may publish the results of this research. However, we will keep your name and other identifying information confidential to the extent allowed by law.

A description of this study will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

# Can I be removed from the research without my OK?

We may remove you from the research study without your approval. Possible reasons for removal would be providing inaccurate answers on the screening survey that affect your eligibility for the study or not following instructions from the researcher during the lab visit.

#### What else do I need to know?

It is not anticipated that participants in this study will experience research-related injury; however, if you need medical care because of taking part in this research study, please contact the investigator to report the issue and contact your primary care physician for medical care. Generally, this care will be billed to you, your insurance, or other third party. Florida State University is not able to offer financial compensation nor to absorb the costs of medical treatment should you be injured as a result of participating in this research.

### Will I be paid for participating in this study?

If you agree to take part in this study, you will be paid up to \$75 in cash for your time and effort: \$10 for the online survey and \$65 for the lab visit. Payment will be distributed after completion of the lab visit.

### Who is funding this study?

This research is being funded by the National Institutes of Health.

# Who can I contact if I have questions about this study?

If you have questions, concerns, or complaints, or think the research has hurt you, talk to the research team:

Dr. Mary A. Gerend, PhD 1105 W. Call Street Florida State University Tallahassee, FL 32306 (850) 645-1541 mary.gerend@med.fsu.edu

This research has been reviewed and approved by the FSU Institutional Review Board ("IRB"). You may talk to them at (850) 644-7900 or humansubjects@fsu.edu if:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You want to talk to someone besides the research team.
- You have questions about your rights as a research subject.
- You want to get information or provide input about this research.

| Do you consent to participate in this study? ☐ Yes ☐ No |
|---|
| To indicate your permission to take part in this research, please type your first and last name below. |

If you would like a copy of this consent form, please print or save a copy of the screen. Alternatively, you can request a copy of the consent form from the experimenter when you are on campus for the lab visit.